CLINICAL TRIAL: NCT03271047
Title: An Open-label Phase 1b/2 Study of Binimetinib Administered in Combination With Nivolumab or Nivolumab Plus Ipilimumab in Patients With Previously Treated Microsatellite-stable (MSS) Metastatic Colorectal Cancer With RAS Mutation
Brief Title: Study of Binimetinib + Nivolumab Plus or Minus Ipilimumab in Patients With Previously Treated Microsatellite-stable (MSS) Metastatic Colorectal Cancer With RAS Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-162-202; C4211004 (Other: Alias Study Number); 2017-003464-12 (EudraCT Number)
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: MSS; RAS-mutant Colorectal Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasms | interventions — binimetinib; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: In phase 1 it is sequential and then in phase 2 it is parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b / Arm 1A (Experimental): binimetinib + nivolumab
  Interventions: Drug: binimetinib; Drug: nivolumab
- Phase 1b / Arm 1B (Experimental): binimetinib + nivolumab + ipilimumab
  Interventions: Drug: binimetinib; Drug: nivolumab; Drug: ipilimumab
- Phase 2 / Arm 2A (Experimental): binimetinib + nivolumab
  Interventions: Drug: binimetinib; Drug: nivolumab
- Phase 2 / Arm 2B (Experimental): binimetinib + nivolumab + ipilimumab
  Interventions: Drug: binimetinib; Drug: nivolumab; Drug: ipilimumab

INTERVENTIONS:
Drug: binimetinib — Orally, twice daily.
Drug: nivolumab — Intravenously (IV) every 4 weeks (Q4W)
Drug: ipilimumab — intravenously (IV) every 8 weeks (Q8W)
  Arms: Phase 1b / Arm 1B; Phase 2 / Arm 2B

SUMMARY:
This is a multicenter, open-label, Phase 1B/2 study to evaluate the safety and assess the preliminary anti-tumor activity of binimetinib administered in combination with nivolumab or nivolumab + ipilimumab in adult patients with advanced metastatic colorectal cancer (mCRC) with microsatellite stable (MSS) disease and presence of a RAS mutation that have received at least one prior line of therapy and no more than 2 prior lines of therapy. The study contains a Phase 1b period to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) and schedule of binimetinib followed by a randomized Phase 2 period to assess the efficacy of the combinations.

ELIGIBILITY:
Key Inclusion Criteria

* Measurable, histologically/cytologically confirmed metastatic colorectal cancer (mCRC).
* Able to provide a sufficient amount of representative tumor specimen for central laboratory testing of RAS mutation status and microsatellite stable (MSS).

  * If a fresh tissue sample is provided, a blood sample is required.
* Metastatic colorectal cancer (mCRC) categorized as microsatellite stable (MSS) by polymerase chain reaction (PCR) per local assay at any time prior to Screening or by the central laboratory.
* RAS mutation per local assay at any time prior to Screening or by the central laboratory.
* Have received at least 1 prior line of therapy and meets at least one of the following criteria:

  * were unable to tolerate the prior first-line regimen
  * experienced disease progression during or after prior first-line regimen for metastatic disease
  * progressed during or within 3 months of completing adjuvant chemotherapy. Note: Generally, treatments that are separated by an event of progression are considered different regimens.
* Have received no more than 2 prior lines of therapy (maintenance therapy given in the metastatic setting will not be considered a separate regimen). Generally, treatments that are separated by an event of progression are considered different regimens.
* Adequate bone marrow, cardiac, kidney and liver function
* Able to take oral medications
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Female patients are either postmenopausal for at least 1 year, are surgically sterile for at least 6 weeks, or must agree to take appropriate precautions to avoid pregnancy from screening through follow-up if of child-bearing potential
* Non-sterile male patients who are sexually active with female partners of childbearing potential must agree to follow instructions for acceptable or highly effective method(s) of contraception for the duration of study treatment and for 7 months after the last dose of study treatment with nivolumab

Key Exclusion Criteria

* Prior treatment with any MEK inhibitor, an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Any untreated central nervous system (CNS) lesion.
* Patients with an active, known or suspected autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Known history of retinal vein occlusion (RVO).
* Known history of Gilbert's syndrome.
* Pregnant or breastfeeding females.
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to first day of study treatment:
* History of thromboembolic or cerebrovascular events ≤ 6 months prior to starting study treatment, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli.
* Uncontrolled hypertension defined as persistent systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy.
* Concurrent neuromuscular disorder that is associated with the potential of elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). NOTE: Testing for HIV must be performed at sites where mandated locally.
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection, and/or detectable virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (33):
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Christiana Care Health Services, Helen F. Graham Cancer Center Pharmacy, Suite 3200, Newark, Delaware
  - Christiana Care Health Services, Helen F. Graham Cancer Center, Newark, Delaware
  - Christiana Care Oncology Hematology, Helen F Graham Cancer Center, Suite 2400, Newark, Delaware
  - Medical Oncology Hematology Consultants, PA, Helen F. Graham Cancer Center, Newark, Delaware
  - Christiana Care Health Services, Christiana Hospital, Newark, Delaware
  - Georgetown University Medical Center Department of Pharmacy, Research, Washington D.C., District of Columbia
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Indiana CTSI Clinical Research Center (ICRC), Indianapolis, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Services IUHSCC, Indianapolis, Indiana
  - Sidney &Lois Eskenazi Hospital, Indianapolis, Indiana
  - Spring Mill Medical Center, Indianapolis, Indiana
  - Siteman Cancer Center - Barnes St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Center for Outpatient Health (Dermatology Clinic), St Louis, Missouri
  - Center for Outpatient Health (Ophthalmology Clinic), St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Investigational Drug Service of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Chattanooga, Tennessee
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Cleveland, Tennessee
  - Tennessee Oncology NASH - SCRI - PPDS, Nashville, Tennessee
  - The Sarah Cannon Research Institute., Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (3):
  - UZ Leuven - Dermatology, Leuven
  - UZ Leuven - Ophthalmology, Leuven
  - UZ Leuven, Leuven
- Netherlands (3):
  - The Netherlands Cancer Institute Antoni Van Leeuwenhoek, Amsterdam, North Holland
  - OLVG locatie Oost, Amsterdam, North Holland
  - Amsterdam Medical Center (AMC), Amsterdam, North Holland
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Rementeria, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital HM Universitario Sanchinarro, CIOCC, Madrid
- United Kingdom (5):
  - Royal Marsden Hospital - London, London, London, CITY of
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Marsden Hospital NHS Foundation Trust, Surrey, Sutton
  - Royal Marsden Hospital NHS Foundation Trust, London
  - Royal Marsden Hospital -Fulham Road, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Elez E, Cubillo A, Alfonso PG, Middleton MR, Chau I, Alkuzweny B, Alcasid A, Zhang X, Van Cutsem E. Binimetinib in combination with nivolumab or nivolumab and ipilimumab in patients with previously treated microsatellite-stable metastatic colorectal cancer with RAS mutations in an open-label phase 1b/2 study. BMC Cancer. 2024 Apr 11;24(1):446. doi: 10.1186/s12885-024-12153-5. PMID 38600471
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-162-202

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included 2 phases: Phase 1b and Phase 2. The recommended dose for Phase 2 (RP2D) of binimetinib was determined in Phase 1b (dose finding phase).
Groups:
- Phase 1b: Nivolumab+Binimetinib: Participants with previously treated microsatellite-stable (MSS) metastatic colorectal cancer with rat sarcoma virus (RAS) mutation received binimetinib at a starting dose of 45 milligrams (mg) tablet orally twice daily (BID) along with 480 mg intravenously (IV) dose of nivolumab every 4 weeks in each 28 day treatment cycle. Binimetinib dose modification to intermitted dosing (3 weeks on treatment and 1 week off treatment) with 45 mg dose or dose reduction to 30 mg BID or 30 mg intermittent dosing based on investigator's decision as per its tolerability among participants. Participants then followed up for safety for around 150 days.
- Phase 1b: Nivolumab+Ipilimumab+Binimetinib: Participants with previously treated MSS metastatic colorectal cancer with RAS mutation received binimetinib at a starting dose of 45 mg tablet BID along with 480 mg IV dose of nivolumab every 4 weeks in each 28 day treatment cycle. Ipilimumab was administered at the dose of 1 milligram per kilogram (mg/kg) IV every 8 weeks after completion of nivolumab infusion. Binimetinib dose modification to intermitted dosing (3 weeks on treatment and 1 week off treatment) with 45 mg dose or dose reduction to 30 mg BID or 30 mg intermittent dosing based on investigator's decision as per its tolerability among participants. Participants then followed up for safety for around 150 days.
- Phase 2: Nivolumab+Binimetinib: Participants with previously treated MSS metastatic colorectal cancer with RAS mutation received 45 mg binimetinib tablet orally BID along with 480 mg IV dose of nivolumab every 4 weeks in each 28 day treatment cycle, until disease progression, unacceptable toxicity, withdrawal of informal consent, initiation of subsequent anticancer therapy, lost to follow-up or death. Participants then followed up for safety for around 150 days.
- Phase 2: Nivolumab+Ipilimumab+Binimetinib: Participants with previously treated MSS metastatic colorectal cancer with RAS mutation received 45 mg binimetinib tablet orally BID along with 480 mg IV dose of nivolumab every 4 weeks in each 28 day treatment cycle. Ipilimumab was administered at the dose of 1 mg/kg IV every 8 weeks after completion of nivolumab infusion until disease progression, unacceptable toxicity, withdrawal of informal consent, initiation of subsequent anticancer therapy, lost to follow-up or death. Participants then followed up for safety for around 150 days.
Period: Phase 1b: Dose Finding Period
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Started | 10 | 11 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 11 | 0 | 0
Not completed — Death | 8 | 8 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Completed follow-up per protocol | 1 | 1 | 0 | 0
Period: Randomized Phase 2 Period
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Started | 0 | 0 | 27 (Participants randomized to Phase 2 of the study.) | 27 (Participants randomized to Phase 2 of the study.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 27 | 27
Not completed — Other | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 20 | 21
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 0
Not completed — Completed follow-up per protocol | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of any study drug in Phase 1b and all participants randomized to study treatment in Phase 2.
Groups:
- Phase 1b: Nivolumab+Binimetinib: Participants with previously treated MSS metastatic colorectal cancer with RAS mutation received binimetinib at a starting dose of 45 mg tablet orally BID along with 480 mg IV dose of nivolumab every 4 weeks in each 28 day treatment cycle. Binimetinib dose modification to intermitted dosing (3 weeks on treatment and 1 week off treatment) with 45 mg dose or dose reduction to 30 mg BID or 30 mg intermittent dosing based on investigator's decision as per its tolerability among participants. Participants then followed up for safety for around 150 days.
- Phase 1b: Nivolumab+Ipilimumab+Binimetinib: Participants with previously treated MSS metastatic colorectal cancer with RAS mutation received binimetinib at a starting dose of 45 mg tablet BID along with 480 mg IV dose of nivolumab every 4 weeks in each 28 day treatment cycle. Ipilimumab was administered at the dose of 1 mg/kg IV every 8 weeks after completion of nivolumab infusion. Binimetinib dose modification to intermitted dosing (3 weeks on treatment and 1 week off treatment) with 45 mg dose or dose reduction to 30 mg BID or 30 mg intermittent dosing based on investigator's decision as per its tolerability among participants. Participants then followed up for safety for around 150 days.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib | Total
Number analyzed (Participants) | 10 | 11 | 27 | 27 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 19 | 20 | 53
  >=65 years | 5 | 2 | 8 | 7 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 11 | 10 | 27
  Male | 8 | 7 | 16 | 17 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 11 | 21 | 23 | 65
  Unknown or Not Reported | 0 | 0 | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 9 | 11 | 21 | 23 | 64
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT:Adverse event(AE)/abnormal laboratory assessed unrelated-disease,disease progression,intercurrent illness/concomitant medication/therapies resulting inability tolerate 75% dose intensity in Cycle 1.Total bilirubin(TBL)grade(G)>=3 (>3.0*upper limit of normal[ULN)]);AST/ALT>5-8*ULN>5 days,>8*ULN,>3*ULN concurrent TBL>2*ULN;G>=3 serum creatinine,CK elevation,ECG QTcF prolonged,G3 troponin,electrolyte>72 hours,G3/4 amylase/lipase.G4 ANC,platelet count>7 days;G3/4 platelet count,other AE except lymphopenia.G>=3 retinopathy,other disorder>21 days;G2 uveitis/eye pain/blurred vision/decreased visual acuity;G4 other disorder.Decrease LVEF>10% G>=3 cardiac disorders.G3/4 hypertension.G3 fatigue>=7 days,hypersensitivity,infusion reaction,fever>=72 hours/hemodynamic compromise,endocrinopathy.G>=2 interstitial lung disease/pneumonitis;G3 bronchospasm.G3/4 rash,hand foot skin reaction,photosensitivity.G3 colitis;G3/4 diarrhea,nausea/vomiting.Neurologic G3.Other hematologic/nonhematolic G>=3 AE.
Time Frame: Cycle 1: Day 1 up to Day 28
Population: Dose-Determining Set (DDS) included all participants in Phase 1b who experienced a DLT or receive at least 75% of the planned binimetinib dose intensity during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 9 | 11
Participants | 1 | 2

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: ORR was defined as the percentage of participants who achieved a best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator per RECIST v1.1. As per RECIST v1.1, CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<)10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-progressive disease (PD). PD was defined as at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was considered progression.
Time Frame: From start of the treatment until disease progression, death or initiation of new anticancer therapy, whichever occurred first (Phase 2: maximum up to 26 months approximately)
Population: All participants randomized to study treatment in Phase 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 27 | 27
Percentage of participants | 0.0 [NA to NA] — Upper and lower limit of 95% confidence interval were not estimable, as there were no participants who had event in this reporting group. | 7.4 [0.9 to 24.3]

3. Secondary Outcome: Phase 1b: Objective Response Rate (ORR) Per RECIST v1.1
Description: ORR was defined as the percentage of participants who achieved a BOR of CR or PR as determined by investigator per RECIST v1.1. As per RECIST v1.1, CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR was defined as at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. Non-target lesions must be non-PD. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From start of the treatment until disease progression, death or initiation of new anticancer therapy, whichever occurred first (Phase 1b: maximum up to 9 months approximately)
Population: All participants who received at least 1 dose of any study treatment in Phase 1b.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11
Percentage of participants | 0.0 [NA to NA] — Upper and lower limit of 95% confidence interval were not estimable, as there were no participants who had event in this reporting group. | 0.0 [NA to NA] — Upper and lower limit of 95% confidence interval were not estimable, as there were no participants who had event in this reporting group.

4. Secondary Outcome: Duration of Response (DOR) as Per RECIST v1.1
Description: DOR was defined as the time between the date of the first documented confirmed response (PR or CR) and the date of the first documented progression or death due to any cause. As per RECIST v1.1: CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes short axis measures <10 mm. PR was defined as at least 30% decrease in sum of measures (tumor lesions- longest diameter and nodes- short axis) of target lesions, taking as reference baseline sum of diameters. PD was defined as at least 20% increase in sum of diameters of measured lesions taking as references smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions.
Time Frame: From date of first documented CR/PR to date of first documented PD, death or initiation of new anticancer therapy, whichever occurred first (Phase 1b: maximum up to 9 months approximately, Phase 2: maximum up to 26 months approximately)
Population: FAS included all participants who received at least 1 dose of any study drug in Phase 1b and all participants randomized to study treatment in Phase 2. Here, "Overall Number of Participants Analyzed" signifies number of participants who achieved an objective response. There were no participants who had event in Phase 1b and Nivolumab and Binimetinib group of Phase 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 0 | 0 | 0 | 2
Months |  |  |  | 11.4 [7.5 to 15.2]

5. Secondary Outcome: Percentage of Participants With Complete Response as Per RECIST v1.1
Description: Complete response as per RECIST v1.1 was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm.
Time Frame: From start of the treatment until disease progression, death or initiation of new anticancer therapy, whichever occurred first (Phase 1b: maximum up to 9 months approximately and Phase 2: maximum up to 26 months approximately)
Population: FAS included all participants who received at least 1 dose of any study drug in Phase 1b and all participants randomized to study treatment in Phase 2.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 27 | 27
Percentage of participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) Based on Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Description: AE: any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE: AE resulting in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs: events between first dose of study drug and up to 30 days after last dose or before start of new anticancer therapy minus 1 day, whichever occurred first. TEAE graded by CTCAE grade 4.03: Grade 3: severe/medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care activities of daily living (ADL); Grade 4: life-threatening consequence, urgent intervention indicated. In this outcome measure, number of participants with 'all grades' and 'Grade 3/4' were reported.
Time Frame: From start of the treatment up to 30 days after last dose or start of new anticancer therapy minus 1 day, whichever occurred first (Phase 1b: maximum up to 9 months approximately and Phase 2: maximum up to 26 months approximately)
Population: The safety set included of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 27 | 27
Participants
  Treatment emergent AEs- All grades | 10 | 11 | 27 | 27
  Treatment emergent SAEs- All grades | 5 | 6 | 12 | 11
  Treatment emergent AEs- Grade 3/4 | 6 | 8 | 19 | 21
  Treatment emergent SAEs- Grade 3/4 | 5 | 6 | 11 | 10

7. Secondary Outcome: Number of Participants With Shift From Baseline in Laboratory Parameter Values Based on Common Terminology Criteria for Adverse Events (CTCAE) v4.03: Hematology and Coagulation
Description: Hematological parameters included: Hemoglobin graded high, Hemoglobin graded low, Platelets count graded low, White Blood Cell (WBC) graded high, WBC graded low, Neutrophils graded low, Lymphocytes graded high, Lymphocytes graded low. Coagulation parameters included: International Normalized Ratio (INR) graded high, Activated Partial Thromboplastin Time (aPTT) graded high. Test abnormalities were graded by CTCAE v4.03 as Grade 1=mild; Grade 2=moderate; Grade 3/Grade 4=severe/life-threatening. A grade 0 was assigned for all non-missing values not graded as 1 or higher. If value was graded >=1 but falls within the normal range, the grade was reset to 0. Categories with at least 1 non-zero data values are reported.
Time Frame: Phase 1b: Baseline up to 30 days after last dose (maximum up to 9 months approximately), Phase 2: Baseline up to 30 days after last dose (maximum up to 26 months approximately)
Population: Safety set included of all participants who received at least 1 dose of study drug. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 27 | 27
Participants
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 7 | 6 | 13 | 16
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 3 | 3 | 4 | 5
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 7 | 6 | 13 | 16
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 2 | 2 | 6 | 10
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 7 | 6 | 13 | 16
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline) | 2 | 1 | 2 | 1
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 7 | 6 | 13 | 16
  Hemoglobin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 1 | 0
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 3 | 5 | 10 | 6
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline) | 0 | 0 | 1 | 0
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 3 | 5 | 10 | 6
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline) | 1 | 4 | 4 | 4
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 3 | 5 | 10 | 6
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline) | 2 | 0 | 3 | 1
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 3 | 5 | 10 | 6
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 3 (at post baseline) | 0 | 1 | 1 | 1
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 3 | 5 | 10 | 6
  Hemoglobin- CTCAE Graded Low: Grade 1 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Hemoglobin- CTCAE Graded Low: Grade 2 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 0 | 4 | 5
  Hemoglobin- CTCAE Graded Low: Grade 2 (at baseline) to Grade 2 (at post baseline) |  |  | 3 | 5
  Hemoglobin- CTCAE Graded Low: Grade 2 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 0 | 4 | 5
  Hemoglobin- CTCAE Graded Low: Grade 2 (at baseline) to Grade 3 (at post baseline) |  |  | 1 | 0
  Hemoglobin- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 10 | 11 | 26 | 26
  Hemoglobin- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 0 | 0 | 1
  Hemoglobin- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 10 | 27 | 27
  Hemoglobin- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Lymphocytes - CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 7 | 9 | 21 | 22
  Lymphocytes - CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 6 | 7 | 11 | 11
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 7 | 9 | 21 | 22
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 0 | 2 | 4
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 7 | 9 | 21 | 22
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 2 | 4 | 6
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 7 | 9 | 21 | 22
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline) | 1 | 0 | 3 | 1
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 7 | 9 | 21 | 22
  Lymphocytes- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Lymphocytes- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1
  Lymphocytes- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline) |  | 0 | 0 | 1
  Lymphocytes- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1
  Lymphocytes- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline) |  | 1 | 1 | 0
  Lymphocytes- CTCAE Graded Low: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1
  Lymphocytes- CTCAE Graded Low: Grade 1 (at baseline) to Grade 3 (at post baseline) |  | 0 | 1 | 0
  Lymphocytes- CTCAE Graded Low: Grade 2 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 2 | 0 | 3 | 4
  Lymphocytes- CTCAE Graded Low: Grade 2 (at baseline) to Grade 0 (at post baseline) | 0 |  | 1 | 0
  Lymphocytes- CTCAE Graded Low: Grade 2 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 2 | 0 | 3 | 4
  Lymphocytes- CTCAE Graded Low: Grade 2 (at baseline) to Grade 2 (at post baseline) | 1 |  | 1 | 2
  Lymphocytes- CTCAE Graded Low: Grade 2 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 2 | 0 | 3 | 4
  Lymphocytes- CTCAE Graded Low: Grade 2 (at baseline) to Grade 3 (at post baseline) | 1 |  | 1 | 2
  Lymphocytes- CTCAE Graded Low: Grade 3 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 1 | 1 | 1 | 0
  Lymphocytes- CTCAE Graded Low: Grade 3 (at baseline) to Grade 0 (at post baseline) | 0 | 0 | 1 |
  Lymphocytes- CTCAE Graded Low: Grade 3 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 1 | 1 | 1 | 0
  Lymphocytes- CTCAE Graded Low: Grade 3 (at baseline) to Grade 2 (at post baseline) | 0 | 1 | 0 |
  Lymphocytes- CTCAE Graded Low: Grade 3 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 1 | 1 | 1 | 0
  Lymphocytes- CTCAE Graded Low: Grade 3 (at baseline) to Grade 3 (at post baseline) | 1 | 0 | 0 |
  Lymphocytes- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 9 | 11 | 25 | 26
  Lymphocytes- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 1 | 0 | 1 | 1
  Lymphocytes- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 11 | 25 | 27
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 9 | 11 | 23 | 26
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 11 | 25 | 27
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 0 | 1 | 1
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 10 | 11 | 25 | 27
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline) | 1 | 0 | 0 | 0
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 25 | 27
  Neutrophils- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Neutrophils- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 2 | 0
  Neutrophils- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline) |  |  | 1 |
  Neutrophils- CTCAE Graded Low: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 0 | 2 | 0
  Neutrophils- CTCAE Graded Low: Grade 1 (at baseline) to Grade 3 (at post baseline) |  |  | 1 |
  Platelets- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 26
  Platelets- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 8 | 9 | 21 | 22
  Platelets- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 26
  Platelets- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 2 | 1 | 3 | 4
  Platelets- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 26
  Platelets- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 2 | 0
  Platelets- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 1 | 1 | 1
  Platelets- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline) |  | 1 | 0 | 0
  Platelets- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 0 | 1 | 1 | 1
  Platelets- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline) |  | 0 | 1 | 1
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 9 | 11 | 21 | 24
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 0 | 2 | 0
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline) | 1 | 0 | 1 | 2
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Grade 4 (at post baseline) | 0 | 0 | 1 | 0
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  WBC- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  WBC- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 1
  WBC- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline) |  |  | 1 | 0
  WBC- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 1
  WBC- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline) |  |  | 0 | 1
  WBC- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 10 | 11 | 26 | 27
  WBC- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  aPTT- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 10 | 24 | 24
  aPTT- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 6 | 8 | 16 | 17
  aPTT- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 10 | 24 | 24
  aPTT- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 3 | 2 | 6 | 6
  aPTT- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 10 | 10 | 24 | 24
  aPTT- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 1 | 0 | 2 | 1
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 1 | 3 | 2
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline) |  | 0 | 0 | 1
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 0 | 1 | 3 | 2
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline) |  | 1 | 1 | 1
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 1 | 3 | 2
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline) |  | 0 | 1 | 0
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 1 | 3 | 2
  aPTT- CTCAE Graded High: Grade 1 (at baseline) to Missing (at post baseline) |  | 0 | 1 | 0
  aPTT- CTCAE Graded High: Missing (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  aPTT- CTCAE Graded High: Missing (at baseline) to Grade 0 (at post baseline) |  |  |  | 1
  INR- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 9 | 8 | 20 | 17
  INR- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 5 | 6 | 16 | 13
  INR- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 9 | 8 | 20 | 17
  INR- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 4 | 2 | 4 | 4
  INR- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 1 | 2 | 7 | 9
  INR- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline) | 0 | 1 | 1 | 1
  INR- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 1 | 2 | 7 | 9
  INR- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline) | 1 | 1 | 5 | 8
  INR- CTCAE Graded High: Grade 1 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 1 | 2 | 7 | 9
  INR- CTCAE Graded High: Grade 1 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  INR- CTCAE Graded High: Grade 2 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0
  INR- CTCAE Graded High: Grade 2 (at baseline) to Grade 2 (at post baseline) |  | 1 |  |
  INR- CTCAE Graded High: Missing (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  INR- CTCAE Graded High: Missing (at baseline) to Grade 0 (at post baseline) |  |  |  | 1

8. Secondary Outcome: Number of Participants With Shift From Baseline in Laboratory Parameter Values Based on Normal Range: Hematology and Coagulation
Description: Hematology parameters: Basophils, Eosinophils, Hematocrit, Monocytes, Red blood cells (RBC). Coagulation parameters: Prothrombin Time. Laboratory values were as per laboratory normal ranges. Values above range were reported as high and values below range as low. Laboratory parameters were graded based on laboratory normal ranges as low, normal, high and missing are reported in this outcome measure. Categories with at least 1 non-zero data values are reported.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 27 | 27
Participants
  Basophils: Normal (at baseline) to Low (at post baseline) | 0 | 0 | 1 | 0
  Basophils: Normal (at baseline) to Normal (at post baseline) | 10 | 11 | 25 | 27
  Basophils: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Eosinophils: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 27
  Eosinophils: Normal (at baseline) to Low (at post baseline) | 0 | 0 | 0 | 1
  Eosinophils: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 27
  Eosinophils: Normal (at baseline) to Normal (at post baseline) | 7 | 11 | 25 | 20
  Eosinophils: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 27
  Eosinophils: Normal (at baseline) to High (at post baseline) | 2 | 0 | 1 | 6
  Eosinophils: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 27
  Eosinophils: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Eosinophils: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 0 | 0 | 0
  Eosinophils: High (at baseline) to Normal (at post baseline) | 1 |  |  |
  Hematocrit: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 2 | 2 | 10 | 9
  Hematocrit: Low (at baseline) to Low (at post baseline) | 2 | 1 | 8 | 9
  Hematocrit: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 2 | 2 | 10 | 9
  Hematocrit: Low (at baseline) to Normal (at post baseline) | 0 | 1 | 1 | 0
  Hematocrit: Low (at baseline) to Missing (at post baseline): number analyzed (Participants) | 2 | 2 | 10 | 9
  Hematocrit: Low (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Hematocrit: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 8 | 9 | 17 | 18
  Hematocrit: Normal (at baseline) to Low (at post baseline) | 5 | 4 | 13 | 12
  Hematocrit: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 8 | 9 | 17 | 18
  Hematocrit: Normal (at baseline) to Normal (at post baseline) | 3 | 4 | 4 | 6
  Hematocrit: Normal (at baseline) to High & Low (at post baseline): number analyzed (Participants) | 8 | 9 | 17 | 18
  Hematocrit: Normal (at baseline) to High & Low (at post baseline) | 0 | 1 | 0 | 0
  Monocytes: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Monocytes: Normal (at baseline) to Low (at post baseline) | 1 | 0 | 1 | 0
  Monocytes: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Monocytes: Normal (at baseline) to Normal (at post baseline) | 9 | 7 | 19 | 20
  Monocytes: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Monocytes: Normal (at baseline) to High (at post baseline) | 0 | 4 | 6 | 6
  Monocytes: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Monocytes: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Monocytes: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  Monocytes: High (at baseline) to Normal (at post baseline) |  |  |  | 1
  RBC: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 1 | 2 | 14 | 7
  RBC: Low (at baseline) to Low (at post baseline) | 1 | 1 | 13 | 6
  RBC: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 2 | 14 | 7
  RBC: Low (at baseline) to Normal (at post baseline) | 0 | 1 | 1 | 1
  RBC: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 8 | 9 | 13 | 19
  RBC: Normal (at baseline) to Low (at post baseline) | 6 | 5 | 8 | 10
  RBC: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 8 | 9 | 13 | 19
  RBC: Normal (at baseline) to Normal (at post baseline) | 2 | 4 | 3 | 9
  RBC: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 8 | 9 | 13 | 19
  RBC: Normal (at baseline) to High (at post baseline) | 0 | 0 | 1 | 0
  RBC: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 8 | 9 | 13 | 19
  RBC: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  RBC: High (at baseline) to Low (at post baseline): number analyzed (Participants) | 1 | 0 | 0 | 1
  RBC: High (at baseline) to Low (at post baseline) | 0 |  |  | 1
  RBC: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 0 | 0 | 1
  RBC: High (at baseline) to Normal (at post baseline) | 1 |  |  | 0
  Prothrombin Time: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 7 | 7 | 19 | 17
  Prothrombin Time: Normal (at baseline) to Normal (at post baseline) | 3 | 3 | 8 | 8
  Prothrombin Time: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 7 | 7 | 19 | 17
  Prothrombin Time: Normal (at baseline) to High (at post baseline) | 4 | 4 | 11 | 9
  Prothrombin Time: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 3 | 4 | 8 | 9
  Prothrombin Time: High (at baseline) to Normal (at post baseline) | 0 | 1 | 0 | 0
  Prothrombin Time: High (at baseline) to High (at post baseline): number analyzed (Participants) | 3 | 4 | 8 | 9
  Prothrombin Time: High (at baseline) to High (at post baseline) | 3 | 3 | 7 | 9
  Prothrombin Time: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 3 | 4 | 8 | 9
  Prothrombin Time: High (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Prothrombin Time: Missing (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  Prothrombin Time: Missing (at baseline) to High (at post baseline) |  |  |  | 1

9. Secondary Outcome: Number of Participants With Shift From Baseline in Laboratory Parameter Values Based on CTCAE v4.03: Chemistry
Description: Abnormalities: Albumin graded low, Alkaline phosphatase (ALP) graded high, Alanine aminotransferase (ALT) graded high, Aspartate aminotransferase (AST) graded high, Bilirubin graded high, Amylase graded high, Creatinine graded high, Corrected calcium graded high, Creatine Kinase (CK) graded high, Glucose graded high, Glucose graded low, Lipase graded high, Magnesium graded high, Magnesium graded low, Potassium graded high, Potassium graded low, Sodium graded high and Sodium graded low. Test abnormalities were graded by CTCAE v4.03 as Grade 1=mild; Grade 2=moderate; Grade 3/Grade 4=severe/life-threatening. A grade 0 was assigned for all non-missing values not graded as 1 or higher. If value was graded >=1 but falls within the normal range, the grade was reset to 0. Categories with at least 1 non-zero data values are reported.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 27 | 27
Participants
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 8 | 10 | 20 | 21
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 5 | 5 | 12 | 12
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 8 | 10 | 20 | 21
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 3 | 5 | 7 | 5
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 8 | 10 | 20 | 21
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 0 | 1 | 1
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 8 | 10 | 20 | 21
  ALT- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 0 | 3
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 1 | 1 | 5 | 5
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline) | 0 | 0 | 1 | 0
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 1 | 1 | 5 | 5
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline) | 1 | 1 | 3 | 2
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 1 | 1 | 5 | 5
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline) | 0 | 0 | 1 | 2
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 1 | 1 | 5 | 5
  ALT- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 0 | 1
  ALT- CTCAE Graded High: Grade 2 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 1 | 0 | 1 | 1
  ALT- CTCAE Graded High: Grade 2 (at baseline) to Grade 2 (at post baseline) | 1 |  | 1 | 0
  ALT- CTCAE Graded High: Grade 2 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 1 | 0 | 1 | 1
  ALT- CTCAE Graded High: Grade 2 (at baseline) to Grade 3 (at post baseline) | 0 |  | 0 | 1
  ALT- CTCAE Graded High: Grade 3 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT- CTCAE Graded High: Grade 3 (at baseline) to Missing (at post baseline) |  |  | 1 |
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 8 | 7 | 21 | 22
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 3 | 2 | 8 | 5
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 8 | 7 | 21 | 22
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 5 | 4 | 11 | 13
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 8 | 7 | 21 | 22
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 1 | 2 | 2
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 8 | 7 | 21 | 22
  AST- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 0 | 2
  AST- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 2 | 4 | 5 | 5
  AST- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline) | 2 | 4 | 3 | 1
  AST- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 2 | 4 | 5 | 5
  AST- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline) | 0 | 0 | 1 | 3
  AST- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 2 | 4 | 5 | 5
  AST- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 1 | 1
  AST- CTCAE Graded High: Grade 2 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 0
  AST- CTCAE Graded High: Grade 2 (at baseline) to Missing (at post baseline) |  |  | 1 |
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 8 | 25 | 26
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 4 | 2 | 8 | 8
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 8 | 25 | 26
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 3 | 2 | 9 | 11
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 10 | 8 | 25 | 26
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline) | 3 | 4 | 7 | 6
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 10 | 8 | 25 | 26
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 0 | 1
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 8 | 25 | 26
  Albumin- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Albumin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 0 | 2 | 2 | 1
  Albumin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline) |  | 0 | 0 | 1
  Albumin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 2 | 2 | 1
  Albumin- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline) |  | 2 | 2 | 0
  Albumin- CTCAE Graded Low: Grade 2 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0
  Albumin- CTCAE Graded Low: Grade 2 (at baseline) to Grade 2 (at post baseline) |  | 1 |  |
  Alkaline phosphatase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 5 | 4 | 15 | 12
  Alkaline phosphatase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 2 | 2 | 7 | 6
  Alkaline phosphatase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 5 | 4 | 15 | 12
  Alkaline phosphatase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 3 | 1 | 8 | 5
  Alkaline phosphatase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 5 | 4 | 15 | 12
  Alkaline phosphatase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 1 | 0 | 1
  Alkaline phosphatase- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 4 | 4 | 9 | 11
  Alkaline phosphatase- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline) | 1 | 0 | 5 | 7
  Alkaline phosphatase- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 4 | 4 | 9 | 11
  Alkaline phosphatase- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline) | 2 | 4 | 3 | 3
  Alkaline phosphatase- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 4 | 4 | 9 | 11
  Alkaline phosphatase- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline) | 1 | 0 | 1 | 1
  Alkaline phosphatase- CTCAE Graded High: Grade 2 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 1 | 1 | 2 | 2
  Alkaline phosphatase- CTCAE Graded High: Grade 2 (at baseline) to Grade 2 (at post baseline) | 0 | 1 | 0 | 0
  Alkaline phosphatase- CTCAE Graded High: Grade 2 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 1 | 1 | 2 | 2
  Alkaline phosphatase- CTCAE Graded High: Grade 2 (at baseline) to Grade 3 (at post baseline) | 1 | 0 | 2 | 2
  Alkaline phosphatase- CTCAE Graded High: Grade 3 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 2 | 1 | 2
  Alkaline phosphatase- CTCAE Graded High: Grade 3 (at baseline) to Grade 3 (at post baseline) |  | 2 | 0 | 2
  Alkaline phosphatase- CTCAE Graded High: Grade 3 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 2 | 1 | 2
  Alkaline phosphatase- CTCAE Graded High: Grade 3 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 26
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 8 | 7 | 18 | 20
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 26
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 1 | 2 | 5 | 2
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 26
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 0 | 1 | 2
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 26
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline) | 0 | 1 | 2 | 2
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 11 | 27 | 26
  Amylase- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 1 | 1 | 0
  Amylase- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 1 | 0 | 0 | 0
  Amylase- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline) | 1 |  |  |
  Amylase- CTCAE Graded High: Grade 2 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  Amylase- CTCAE Graded High: Grade 2 (at baseline) to Grade 4 (at post baseline) |  |  |  | 1
  Bilirubin- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 27
  Bilirubin- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 10 | 9 | 25 | 24
  Bilirubin- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 27
  Bilirubin- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 0 | 1 | 2
  Bilirubin- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 27
  Bilirubin- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 1 | 0 | 1
  Bilirubin- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0
  Bilirubin- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline) |  | 1 |  |
  Bilirubin- CTCAE Graded High: Grade 4 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 0
  Bilirubin- CTCAE Graded High: Grade 4 (at baseline) to Missing (at post baseline) |  |  | 1 |
  Corrected Calcium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Corrected Calcium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 7 | 11 | 24 | 25
  Corrected Calcium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Corrected Calcium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 3 | 0 | 2 | 1
  Corrected Calcium- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Corrected Calcium- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Corrected Calcium- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  Corrected Calcium- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline) |  |  |  | 1
  Corrected Calcium- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Corrected Calcium- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 10 | 11 | 25 | 25
  Corrected Calcium- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Corrected Calcium- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 0 | 1 | 1
  Corrected Calcium- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 27 | 26
  Corrected Calcium- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Corrected Calcium- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  Corrected Calcium- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline) |  |  |  | 1
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 9 | 10 | 27 | 23
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 1 | 3 | 3 | 7
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 9 | 10 | 27 | 23
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 3 | 4 | 11 | 7
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 9 | 10 | 27 | 23
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 4 | 2 | 6 | 8
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 9 | 10 | 27 | 23
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline) | 1 | 1 | 5 | 1
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 9 | 10 | 27 | 23
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Grade 4 (at post baseline) | 0 | 0 | 1 | 0
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 10 | 27 | 23
  Creatine kinase- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Creatine kinase- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 1 | 1 | 0 | 3
  Creatine kinase- CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline) | 0 | 1 |  | 1
  Creatine kinase- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 1 | 1 | 0 | 3
  Creatine kinase- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline) | 1 | 0 |  | 1
  Creatine kinase- CTCAE Graded High: Grade 1 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 1 | 1 | 0 | 3
  Creatine kinase- CTCAE Graded High: Grade 1 (at baseline) to Grade 4 (at post baseline) | 0 | 0 |  | 1
  Creatine kinase - CTCAE Graded High: Missing (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  Creatine kinase - CTCAE Graded High: Missing (at baseline) to Grade 1 (at post baseline) |  |  |  | 1
  Creatinine- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 1 | 2 | 6 | 7
  Creatinine- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 7 | 7 | 14 | 18
  Creatinine- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 2 | 2 | 5 | 2
  Creatinine- CTCAE Graded High: Grade 0 (at baseline) to Grade 4 (at post baseline) | 0 | 0 | 1 | 0
  Creatinine- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 10 | 10 | 23 | 26
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 1 | 1 | 0
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 0 | 1 | 0
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 26
  Glucose- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Glucose- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 1
  Glucose- CTCAE Graded Low: Grade 1 (at baseline) to Grade 0 (at post baseline) |  |  | 0 | 1
  Glucose- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 1
  Glucose- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline) |  |  | 1 | 0
  Glucose- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 9 | 10 | 24 | 21
  Glucose- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 7 | 6 | 18 | 14
  Glucose- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 9 | 10 | 24 | 21
  Glucose- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 1 | 1 | 1
  Glucose - CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 9 | 10 | 24 | 21
  Glucose - CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 1 | 1 | 0 | 1
  Glucose- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 10 | 24 | 21
  Glucose- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 1 | 2 | 5 | 5
  Glucose- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 1
  Glucose- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline) |  |  | 1 | 0
  Glucose - CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 1
  Glucose - CTCAE Graded High: Grade 1 (at baseline) to Grade 2 (at post baseline) |  |  | 0 | 1
  Glucose- CTCAE Graded High: Grade 3 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 2
  Glucose- CTCAE Graded High: Grade 3 (at baseline) to Grade 2 (at post baseline) |  |  | 1 | 0
  Glucose- CTCAE Graded High: Grade 3 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 2
  Glucose- CTCAE Graded High: Grade 3 (at baseline) to Grade 3 (at post baseline) |  |  | 0 | 1
  Glucose- CTCAE Graded High: Grade 3 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 2
  Glucose- CTCAE Graded High: Grade 3 (at baseline) to Missing (at post baseline) |  |  | 0 | 1
  Glucose- CTCAE Graded High: Missing (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 1 | 1 | 1 | 3
  Glucose- CTCAE Graded High: Missing (at baseline) to Grade 0 (at post baseline) | 0 | 0 | 0 | 1
  Glucose- CTCAE Graded High: Missing (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 1 | 1 | 1 | 3
  Glucose- CTCAE Graded High: Missing (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 1 | 0
  Glucose- CTCAE Graded High: Missing (at baseline) to Missing (at post baseline): number analyzed (Participants) | 1 | 1 | 1 | 3
  Glucose- CTCAE Graded High: Missing (at baseline) to Missing (at post baseline) | 1 | 1 | 0 | 2
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 9 | 10 | 25 | 23
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 5 | 6 | 17 | 15
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 9 | 10 | 25 | 23
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 2 | 2 | 2 | 4
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 9 | 10 | 25 | 23
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 2 (at post baseline) | 1 | 1 | 1 | 0
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 9 | 10 | 25 | 23
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 3 (at post baseline) | 1 | 0 | 4 | 3
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 9 | 10 | 25 | 23
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Grade 4 (at post baseline) | 0 | 0 | 0 | 1
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 10 | 25 | 23
  Lipase- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 1 | 1 | 0
  Lipase- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 1 | 1 | 2 | 3
  Lipase- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline) | 1 | 0 | 1 | 0
  Lipase- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 1 | 1 | 2 | 3
  Lipase- CTCAE Graded High: Grade 1 (at baseline) to Grade 1 (at post baseline) | 0 | 1 | 1 | 2
  Lipase- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 1 | 1 | 2 | 3
  Lipase- CTCAE Graded High: Grade 1 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 0 | 1
  Lipase- CTCAE Graded High: Grade 4 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  Lipase- CTCAE Graded High: Grade 4 (at baseline) to Grade 4 (at post baseline) |  |  |  | 1
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 9 | 11 | 26 | 27
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 8 | 10 | 22 | 24
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 9 | 11 | 26 | 27
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 1 | 1 | 3 | 2
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 9 | 11 | 26 | 27
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 2 (at post baseline) | 0 | 0 | 0 | 1
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 11 | 26 | 27
  Magnesium- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Magnesium- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline): number analyzed (Participants) | 1 | 0 | 0 | 0
  Magnesium- CTCAE Graded Low: Grade 1 (at baseline) to Grade 2 (at post baseline) | 1 |  |  |
  Magnesium- CTCAE Graded Low: Grade 2 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 0
  Magnesium- CTCAE Graded Low: Grade 2 (at baseline) to Grade 3 (at post baseline) |  |  | 1 |
  Magnesium- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 10 | 11 | 26 | 27
  Magnesium- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 7 | 9 | 20 | 23
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 3 | 2 | 3 | 4
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 1 | 0
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 4 (at post baseline) | 0 | 0 | 1 | 0
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded Low: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Potassium- CTCAE Graded Low: Grade 3 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium- CTCAE Graded Low: Grade 3 (at baseline) to Grade 3 (at post baseline) |  |  | 1 |
  Potassium- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 9 | 10 | 23 | 23
  Potassium- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 1 | 1 | 2 | 4
  Potassium- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 27
  Potassium- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Potassium- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium- CTCAE Graded High: Grade 1 (at baseline) to Grade 0 (at post baseline) |  |  | 1 |
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 27
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 0 (at post baseline) | 9 | 7 | 19 | 23
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 27
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 1 (at post baseline) | 1 | 3 | 3 | 1
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 27
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 3 (at post baseline) | 0 | 0 | 1 | 2
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 4 (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 27
  Sodium- CTCAE Graded Low: Grade 0 (at baseline) to Grade 4 (at post baseline) | 0 | 0 | 2 | 1
  Sodium- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline): number analyzed (Participants) | 0 | 0 | 2 | 0
  Sodium- CTCAE Graded Low: Grade 1 (at baseline) to Grade 1 (at post baseline) |  |  | 1 |
  Sodium- CTCAE Graded Low: Grade 1 (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 0 | 2 | 0
  Sodium- CTCAE Graded Low: Grade 1 (at baseline) to Missing (at post baseline) |  |  | 1 |
  Sodium- CTCAE Graded Low: Grade 3 (at baseline) to Grade 3 (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0
  Sodium- CTCAE Graded Low: Grade 3 (at baseline) to Grade 3 (at post baseline) |  | 1 |  |
  Sodium- CTCAE Graded High: Grade 0 (at baseline) to Grade 0 (at post baseline) | 10 | 11 | 23 | 22
  Sodium- CTCAE Graded High: Grade 0 (at baseline) to Grade 1 (at post baseline) | 0 | 0 | 3 | 5
  Sodium- CTCAE Graded High: Grade 0 (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0

10. Secondary Outcome: Number of Participants With Shift From Baseline in Laboratory Parameter Values Based on Normal Range: Chemistry and Thyroid Function
Description: Chemistry laboratory parameters: Blood urea nitrogen (BUN), Total protein, Chloride, Cancer antigen 19-9 (CA 19-9), Brain natriuretic peptide (BNP), Bicarbonate, Direct bilirubin, Carcinoembryonic antigen (CEA), Lactate dehydrogenase (LDH), Uric acid, Troponin I. Thyroid panel laboratory parameters: Thyroid-stimulating hormone (TSH), Free triiodothyronine (T3), Free thyroxine (T4). Laboratory values were as per laboratory normal ranges. Values above range were reported as high and values below range as low. Shift in chemistry and thyroid panel severity from baseline grade low, normal, high and missing to the post baseline grades as low, normal, high and missing are reported in this outcome measure. Categories with at least 1 non-zero data values are reported.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 27 | 27
Participants
  BNP: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 9 | 9 | 27 | 25
  BNP: Normal (at baseline) to Normal (at post baseline) | 8 | 6 | 24 | 22
  BNP: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 9 | 9 | 27 | 25
  BNP: Normal (at baseline) to High (at post baseline) | 1 | 3 | 2 | 3
  BNP: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 9 | 27 | 25
  BNP: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  BNP: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 2 | 0 | 2
  BNP: High (at baseline) to Normal (at post baseline) | 0 | 2 |  | 0
  BNP: High (at baseline) to High (at post baseline): number analyzed (Participants) | 1 | 2 | 0 | 2
  BNP: High (at baseline) to High (at post baseline) | 1 | 0 |  | 2
  BUN: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 7 | 9 | 25 | 21
  BUN: Normal (at baseline) to Normal (at post baseline) | 4 | 3 | 15 | 14
  BUN (mmol/L): Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 7 | 9 | 25 | 21
  BUN (mmol/L): Normal (at baseline) to High (at post baseline) | 3 | 5 | 9 | 7
  BUN: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 7 | 9 | 25 | 21
  BUN: Normal (at baseline) to Missing (at post baseline) | 0 | 1 | 1 | 0
  BUN: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 3 | 2 | 2 | 6
  BUN: High (at baseline) to Normal (at post baseline) | 0 | 0 | 2 | 3
  BUN: High (at baseline) to High (at post baseline): number analyzed (Participants) | 3 | 2 | 2 | 6
  BUN: High (at baseline) to High (at post baseline) | 3 | 2 | 0 | 3
  Bicarbonate: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 2 | 1 | 3
  Bicarbonate: Low (at baseline) to Normal (at post baseline) |  | 1 | 0 | 3
  Bicarbonate: Low (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 2 | 1 | 3
  Bicarbonate: Low (at baseline) to High (at post baseline) |  | 1 | 1 | 0
  Bicarbonate: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 10 | 9 | 26 | 24
  Bicarbonate: Normal (at baseline) to Low (at post baseline) | 2 | 1 | 6 | 9
  Bicarbonate: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 10 | 9 | 26 | 24
  Bicarbonate: Normal (at baseline) to Normal (at post baseline) | 7 | 6 | 18 | 11
  Bicarbonate: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 10 | 9 | 26 | 24
  Bicarbonate: Normal (at baseline) to High (at post baseline) | 1 | 2 | 1 | 3
  Bicarbonate: Normal (at baseline) to High and Low (at post baseline): number analyzed (Participants) | 10 | 9 | 26 | 24
  Bicarbonate: Normal (at baseline) to High and Low (at post baseline) | 0 | 0 | 0 | 1
  Bicarbonate: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 9 | 26 | 24
  Bicarbonate: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  CA 19-9: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 3 | 4 | 8 | 9
  CA 19-9: Normal (at baseline) to Normal (at post baseline) | 3 | 3 | 6 | 7
  CA 19-9: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 3 | 4 | 8 | 9
  CA 19-9: Normal (at baseline) to High (at post baseline) | 0 | 0 | 2 | 1
  CA 19-9: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 3 | 4 | 8 | 9
  CA 19-9: Normal (at baseline) to Missing (at post baseline) | 0 | 1 | 0 | 1
  CA 19-9: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 7 | 7 | 19 | 18
  CA 19-9: High (at baseline) to Normal (at post baseline) | 0 | 0 | 1 | 1
  CA 19-9: High (at baseline) to High (at post baseline): number analyzed (Participants) | 7 | 7 | 19 | 18
  CA 19-9: High (at baseline) to High (at post baseline) | 7 | 6 | 16 | 16
  CA 19-9: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 7 | 7 | 19 | 18
  CA 19-9: High (at baseline) to Missing (at post baseline) | 0 | 1 | 2 | 1
  CEA: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 0 | 3 | 6
  CEA: Normal (at baseline) to Normal (at post baseline) | 1 |  | 1 | 3
  CEA: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 1 | 0 | 3 | 6
  CEA: Normal (at baseline) to High (at post baseline) | 0 |  | 2 | 2
  CEA: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 1 | 0 | 3 | 6
  CEA: Normal (at baseline) to Missing (at post baseline) | 0 |  | 0 | 1
  CEA: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 9 | 11 | 24 | 21
  CEA: High (at baseline) to Normal (at post baseline) | 0 | 0 | 1 | 0
  CEA: High (at baseline) to High (at post baseline): number analyzed (Participants) | 9 | 11 | 24 | 21
  CEA: High (at baseline) to High (at post baseline) | 9 | 9 | 20 | 20
  CEA: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 11 | 24 | 21
  CEA: High (at baseline) to Missing (at post baseline) | 0 | 2 | 3 | 1
  Chloride: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1
  Chloride: Low (at baseline) to Low (at post baseline) |  | 1 | 1 | 1
  Chloride: Low (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1
  Chloride: Low (at baseline) to Missing (at post baseline) |  | 0 | 1 | 0
  Chloride: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 26
  Chloride: Normal (at baseline) to Low (at post baseline) | 2 | 2 | 8 | 3
  Chloride: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 26
  Chloride: Normal (at baseline) to Normal (at post baseline) | 8 | 7 | 15 | 22
  Chloride: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 26
  Chloride: Normal (at baseline) to High (at post baseline) | 0 | 0 | 2 | 1
  Chloride: Normal (at baseline) to High & Low (at post baseline): number analyzed (Participants) | 10 | 10 | 25 | 26
  Chloride: Normal (at baseline) to High & Low (at post baseline) | 0 | 1 | 0 | 0
  Free T3: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 2
  Free T3: Low (at baseline) to Low (at post baseline) |  |  | 0 | 1
  Free T3: Low (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 2
  Free T3: Low (at baseline) to Missing (at post baseline) |  |  | 1 | 1
  Free T3: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 23
  Free T3: Normal (at baseline) to Low (at post baseline) | 3 | 5 | 8 | 7
  Free T3: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 23
  Free T3: Normal (at baseline) to Normal (at post baseline) | 7 | 5 | 15 | 15
  Free T3: Normal (at baseline) to High and Low (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 23
  Free T3: Normal (at baseline) to High and Low (at post baseline) | 0 | 0 | 1 | 0
  Free T3: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 11 | 26 | 23
  Free T3: Normal (at baseline) to Missing (at post baseline) | 0 | 1 | 2 | 1
  Free T3: High (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 2
  Free T3: High (at baseline) to High (at post baseline) |  |  |  | 2
  Free T4: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 1
  Free T4: Low (at baseline) to Low (at post baseline) |  | 0 |  | 1
  Free T4: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 1
  Free T4: Low (at baseline) to Normal (at post baseline) |  | 1 |  | 0
  Free T4: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 24
  Free T4: Normal (at baseline) to Low (at post baseline) | 0 | 1 | 2 | 3
  Free T4: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 24
  Free T4: Normal (at baseline) to Normal (at post baseline) | 10 | 8 | 17 | 17
  Free T4: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 24
  Free T4: Normal (at baseline) to High (at post baseline) | 0 | 0 | 3 | 1
  Free T4: Normal (at baseline) to High and Low (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 24
  Free T4: Normal (at baseline) to High and Low (at post baseline) | 0 | 0 | 1 | 1
  Free T4: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 10 | 26 | 24
  Free T4: Normal (at baseline) to Missing (at post baseline) | 0 | 1 | 3 | 2
  Free T4: High (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 2
  Free T4: High (at baseline) to Low (at post baseline) |  |  | 0 | 1
  Free T4: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 0 | 1 | 2
  Free T4: High (at baseline) to Normal (at post baseline) |  |  | 1 | 1
  LDH: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 1 | 0 | 0 | 0
  LDH: Low (at baseline) to Low (at post baseline) | 1 |  |  |
  LDH: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 6 | 5 | 20 | 15
  LDH: Normal (at baseline) to Normal (at post baseline) | 1 | 1 | 6 | 5
  LDH: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 6 | 5 | 20 | 15
  LDH: Normal (at baseline) to High (at post baseline) | 5 | 4 | 14 | 10
  LDH: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 3 | 6 | 7 | 12
  LDH: High (at baseline) to Normal (at post baseline) | 0 | 0 | 0 | 1
  LDH: High (at baseline) to High (at post baseline): number analyzed (Participants) | 3 | 6 | 7 | 12
  LDH: High (at baseline) to High (at post baseline) | 3 | 6 | 6 | 11
  LDH: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 3 | 6 | 7 | 12
  LDH: High (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  Protein: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0
  Protein: Low (at baseline) to Low (at post baseline) |  | 1 |  |
  Protein: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 10 | 10 | 27 | 27
  Protein: Normal (at baseline) to Low (at post baseline) | 5 | 6 | 11 | 11
  Protein: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 10 | 10 | 27 | 27
  Protein: Normal (at baseline) to Normal (at post baseline) | 5 | 4 | 12 | 14
  Protein: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 10 | 10 | 27 | 27
  Protein: Normal (at baseline) to High (at post baseline) | 0 | 0 | 0 | 2
  Protein: Normal (at baseline) to High and Low (at post baseline): number analyzed (Participants) | 10 | 10 | 27 | 27
  Protein: Normal (at baseline) to High and Low (at post baseline) | 0 | 0 | 3 | 0
  Protein: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 10 | 10 | 27 | 27
  Protein: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 1 | 0
  TSH: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1
  TSH: Low (at baseline) to Low (at post baseline) |  |  |  | 1
  TSH: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 9 | 7 | 24 | 26
  TSH: Normal (at baseline) to Low (at post baseline) | 0 | 0 | 2 | 3
  TSH: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 9 | 7 | 24 | 26
  TSH: Normal (at baseline) to Normal (at post baseline) | 8 | 7 | 14 | 20
  TSH: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 9 | 7 | 24 | 26
  TSH: Normal (at baseline) to High (at post baseline) | 1 | 0 | 3 | 1
  TSH: Normal (at baseline) to High and Low (at post baseline): number analyzed (Participants) | 9 | 7 | 24 | 26
  TSH: Normal (at baseline) to High and Low (at post baseline) | 0 | 0 | 2 | 0
  TSH: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 9 | 7 | 24 | 26
  TSH: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 3 | 2
  TSH: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 4 | 3 | 0
  TSH: High (at baseline) to Normal (at post baseline) | 0 | 2 | 2 |
  TSH: High (at baseline) to High (at post baseline): number analyzed (Participants) | 1 | 4 | 3 | 0
  TSH: High (at baseline) to High (at post baseline) | 1 | 1 | 1 |
  TSH: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 1 | 4 | 3 | 0
  TSH: High (at baseline) to Missing (at post baseline) | 0 | 1 | 0 |
  Troponin I: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 2 | 26 | 26
  Troponin I: Normal (at baseline) to Normal (at post baseline) |  | 2 | 11 | 10
  Troponin I: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 2 | 26 | 26
  Troponin I: Normal (at baseline) to High (at post baseline) |  | 0 | 1 | 2
  Troponin I: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 2 | 26 | 26
  Troponin I: Normal (at baseline) to Missing (at post baseline) |  | 0 | 14 | 14
  Troponin I: Missing (at baseline) to Normal (at post baseline): number analyzed (Participants) | 5 | 3 | 0 | 1
  Troponin I: Missing (at baseline) to Normal (at post baseline) | 4 | 3 |  | 1
  Troponin I: Missing (at baseline) to High (at post baseline): number analyzed (Participants) | 5 | 3 | 0 | 1
  Troponin I: Missing (at baseline) to High (at post baseline) | 1 | 0 |  | 0
  Uric acid: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 1 | 1 | 3
  Uric acid: Low (at baseline) to Low (at post baseline) |  | 0 | 0 | 2
  Uric acid: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 1 | 1 | 3
  Uric acid: Low (at baseline) to Normal (at post baseline) |  | 1 | 0 | 1
  Uric acid: Low (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 1 | 1 | 3
  Uric acid: Low (at baseline) to Missing (at post baseline) |  | 0 | 1 | 0
  Uric acid: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 9 | 9 | 23 | 21
  Uric acid: Normal (at baseline) to Low (at post baseline) | 1 | 2 | 4 | 4
  Uric acid: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 9 | 9 | 23 | 21
  Uric acid: Normal (at baseline) to Normal (at post baseline) | 8 | 5 | 15 | 16
  Uric acid: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 9 | 9 | 23 | 21
  Uric acid: Normal (at baseline) to High (at post baseline) | 0 | 2 | 4 | 1
  Uric acid: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 1 | 3 | 3
  Uric acid: High (at baseline) to Normal (at post baseline) | 0 | 0 | 1 | 0
  Uric acid: High (at baseline) to High (at post baseline): number analyzed (Participants) | 1 | 1 | 3 | 3
  Uric acid: High (at baseline) to High (at post baseline) | 1 | 1 | 2 | 3

11. Secondary Outcome: Number of Participants With Abnormal Hepatic Laboratory Values
Description: Criteria for abnormal hepatic laboratory parameters: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT): >3* upper limit of normal (ULN), >5*ULN, >8*ULN, >10*ULN, >20*ULN; Total bilirubin (TBL) >1.5*ULN, >2*ULN; Alkaline phosphatase (ALP) >2*ULN, >3*ULN. Categories with at least 1 non-zero data values are reported.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 27 | 27
Participants
  ALT: >3 ULN: number analyzed (Participants) | 9 | 11 | 25 | 26
  ALT: >3 ULN | 0 | 0 | 2 | 7
  ALT: >5 ULN: number analyzed (Participants) | 10 | 11 | 26 | 27
  ALT: >5 ULN | 0 | 0 | 0 | 5
  ALT: >8 ULN: number analyzed (Participants) | 10 | 11 | 26 | 27
  ALT: >8 ULN | 0 | 0 | 0 | 1
  AST: >3 ULN: number analyzed (Participants) | 10 | 11 | 26 | 27
  AST: >3 ULN | 0 | 1 | 4 | 8
  AST: >5 ULN: number analyzed (Participants) | 10 | 11 | 26 | 27
  AST: >5 ULN | 0 | 0 | 1 | 3
  AST: >8 ULN: number analyzed (Participants) | 10 | 11 | 26 | 27
  AST: >8 ULN | 0 | 0 | 1 | 1
  ALT or AST: >3 ULN: number analyzed (Participants) | 9 | 11 | 25 | 26
  ALT or AST: >3 ULN | 0 | 1 | 3 | 7
  ALT or AST: >5 ULN: number analyzed (Participants) | 10 | 11 | 26 | 27
  ALT or AST: >5 ULN | 0 | 0 | 1 | 4
  ALT or AST: >8 ULN: number analyzed (Participants) | 10 | 11 | 26 | 27
  ALT or AST: >8 ULN | 0 | 0 | 1 | 1
  Total bilirubin: >1.5 ULN: number analyzed (Participants) | 9 | 11 | 26 | 26
  Total bilirubin: >1.5 ULN | 0 | 2 | 0 | 1
  Alkaline phosphatase: >2 ULN: number analyzed (Participants) | 8 | 6 | 22 | 22
  Alkaline phosphatase: >2 ULN | 3 | 3 | 4 | 8
  Alkaline phosphatase: >3 ULN: number analyzed (Participants) | 10 | 8 | 24 | 24
  Alkaline phosphatase: >3 ULN | 4 | 4 | 2 | 4

12. Secondary Outcome: Concentration Versus Time Summary of Plasma Concentration of Binimetinib
Time Frame: 1.5 hours post dose of binimetinib on Day 1, 15 of Cycle 1; pre dose of binimetinib on Day 15 of Cycle 1, 2, 3, 4, 5
Population: The pharmacokinetic analysis set included of all participants who received at least 1 dose of binimetinib and have at least one evaluable bioanalytical result. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
Number analyzed (Participants) | 10 | 11 | 26 | 27
nanogram per milliliter
  Cycle 1 Day 1: 1.5 Hours post dose: number analyzed (Participants) | 10 | 11 | 21 | 23
  Cycle 1 Day 1: 1.5 Hours post dose | 228 (152.2) | 163 (129.6) | 261 (90.9) | 217 (134.5)
  Cycle 1 Day 15: pre dose: number analyzed (Participants) | 4 | 5 | 12 | 8
  Cycle 1 Day 15: pre dose | 135 (60.9) | 125 (103.9) | 77.0 (141.2) | 81.8 (143.6)
  Cycle 1 Day 15: 1.5 Hours post dose: number analyzed (Participants) | 4 | 8 | 15 | 18
  Cycle 1 Day 15: 1.5 Hours post dose | 542 (57.6) | 414 (24.5) | 294 (84.4) | 324 (83.3)
  Cycle 2 Day 15: pre dose: number analyzed (Participants) | 4 | 2 | 7 | 7
  Cycle 2 Day 15: pre dose | 108 (52.9) | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below the limit of quantification (LOQ). | 88.5 (111.3) | 120 (77.7)
  Cycle 3 Day 15: pre dose: number analyzed (Participants) | 3 | 2 | 1 | 3
  Cycle 3 Day 15: pre dose | 140 (42.0) | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ. | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ. | 89.2 (183.4)
  Cycle 4 Day 15: pre dose: number analyzed (Participants) | 2 | 1 | 1 | 1
  Cycle 4 Day 15: pre dose | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ. | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ. | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ. | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ.
  Cycle 5 Day 15: pre dose: number analyzed (Participants) | 1 | 0 | 1 | 1
  Cycle 5 Day 15: pre dose | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ. |  | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ. | NA (NA) — Geometric mean and geometric coefficient of variation were not estimable as concentration was below LOQ.

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From start of the treatment up to 150 days after last dose (Phase 1b: maximum up to 13 months approximately and Phase 2: maximum up to 30 months approximately); TEAEs (including serious and other AEs): From start of the treatment up to 30 days after last dose (Phase 1b: maximum up to 9 months approximately and Phase 2: maximum up to 26 months approximately)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety set was evaluated. Both TEAE and treatment related AEs were monitored.
Arm/Group | Phase 1b: Nivolumab+Binimetinib | Phase 1b: Nivolumab+Ipilimumab+Binimetinib | Phase 2: Nivolumab+Binimetinib | Phase 2: Nivolumab+Ipilimumab+Binimetinib
All-Cause Mortality (participants affected / at risk) | 8/10 | 8/11 | 20/27 | 21/27
Serious Adverse Events (participants affected / at risk) | 5/10 | 6/11 | 12/27 | 11/27
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11 | 27/27 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Nivolumab+Binimetinib (N=10) | Phase 1b: Nivolumab+Ipilimumab+Binimetinib (N=11) | Phase 2: Nivolumab+Binimetinib (N=27) | Phase 2: Nivolumab+Ipilimumab+Binimetinib (N=27)
Myocarditis (Cardiac disorders) | 0 | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 1
Infected seroma (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Nivolumab+Binimetinib (N=10) | Phase 1b: Nivolumab+Ipilimumab+Binimetinib (N=11) | Phase 2: Nivolumab+Binimetinib (N=27) | Phase 2: Nivolumab+Ipilimumab+Binimetinib (N=27)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 7 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 1
Visual impairment (Eye disorders) | 2 | 1 | 0 | 3
Periorbital oedema (Eye disorders) | 1 | 0 | 3 | 1
Vision blurred (Eye disorders) | 1 | 1 | 1 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 2
Subretinal fluid (Eye disorders) | 0 | 0 | 2 | 1
Macular oedema (Eye disorders) | 0 | 0 | 2 | 0
Photopsia (Eye disorders) | 0 | 1 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 0 | 2
Dry age-related macular degeneration (Eye disorders) | 1 | 0 | 0 | 0
Eye oedema (Eye disorders) | 1 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 13 | 15
Nausea (Gastrointestinal disorders) | 5 | 2 | 12 | 11
Vomiting (Gastrointestinal disorders) | 2 | 8 | 7 | 10
Constipation (Gastrointestinal disorders) | 2 | 3 | 9 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 5 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 3 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 5
Ascites (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 6 | 11 | 11
Oedema peripheral (General disorders) | 5 | 5 | 8 | 11
Pyrexia (General disorders) | 3 | 3 | 8 | 14
Asthenia (General disorders) | 3 | 1 | 7 | 9
Chills (General disorders) | 1 | 1 | 4 | 4
Face oedema (General disorders) | 0 | 1 | 4 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 3
Influenza like illness (General disorders) | 0 | 2 | 1 | 0
Paronychia (Infections and infestations) | 1 | 1 | 3 | 3
Rash pustular (Infections and infestations) | 1 | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 5 | 3 | 14 | 13
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 2 | 9
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2 | 8
Ejection fraction decreased (Investigations) | 1 | 0 | 4 | 7
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 5
Amylase increased (Investigations) | 0 | 0 | 3 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 2
Lipase increased (Investigations) | 0 | 0 | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 2
Troponin T increased (Investigations) | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 1 | 2
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0
Troponin I increased (Investigations) | 1 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 13 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal colic (Renal and urinary disorders) | 0 | 1 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 6 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 6 | 13 | 12
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 8 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 5 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 3 | 4
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT03271047/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03271047/SAP_001.pdf